CLINICAL TRIAL: NCT04030364
Title: Implementation of a Multi-component, Supervised Exercise Program for Patients With Type 2 Diabetes Mellitus From a Primary Care Practice: A Quality Improvement Study.
Brief Title: Implementation of a Multi-component, Supervised Exercise Program for Patients With Type 2 Diabetes Mellitus.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190116-01H
Record Dates: First submitted 2019-07-05; First posted 2019-07-24 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-referral to group exercise classes (Other): Structured, multi-component, supervised group exercise classes are the health related intervention proposed for this study. The group classes will occur at a local CrossFit gym facility.
  For the purposes of this project, all eligible Rosemount Clinic patients with type 2 diabetes mellitus will receive an email or letter mail invitation to self-refer to a structured, facility-based, supervised aerobic and resistance exercise program. Interested patients will be invited to attend a 1-hour information session at the exercise facility at the time of implementation start up where they will complete an initial baseline survey. This session will also serve as an initial meet and greet for participants to meet exercise trainers prior to starting exercise classes and to receive a tour of the facility.
  Interventions: Behavioral: CrossFit group exercise classes

INTERVENTIONS:
Behavioral: CrossFit group exercise classes — The group classes will occur at a local CrossFit gym facility. Participants will be free to attend up to 6 regularly-scheduled, free, 1-hr group classes per week at the local exercise facility for a period of 3-months. The recommendation will be to aim to attend at least three classes/week but there will no prescribed minimum. Classes will be supervised by experienced trainers.
  Trainers will work collaboratively with participants to adapt the skill and workout of the day within each group class to the individual participant's physical limitations and needs. As such, each participant may complete a slightly different movement or workout on any given day based on their functional status at that time. However, all participants will be actively included in the community of the group class and will experience a relative stimulus that is moderately challenging for them.

SUMMARY:
This quality improvement study aims to implement a supervised, multi-component exercise program for patients type 2 diabetes mellitus (T2DM) from a primary care practice. Rosemount Clinic patients with T2DM will be invited to participate in free group exercise classes as part of a 3-month program of structured exercise to enhance adherence to the Canadian Diabetes Association (CDA) clinical best practice guidelines. Interested patients will attend an initial 1-hour information session and then will complete short, monthly questionnaires about their current quality of life and experience with the exercise program. Participation is voluntary and patients may drop out at any time.

DETAILED DESCRIPTION:
The Canadian Diabetes Association 2018 Clinical Practice Guidelines state that moderate to high levels of physical activity and cardiorespiratory fitness are associated with substantially lower morbidity and mortality in people with diabetes. The recommendations include a combination of aerobic, resistance, and flexibility exercises. The Guidelines specifically advocate for strategies that increase self-efficacy and motivation in order to increase physical activity uptake and maintenance.

Similarly, the importance of exercise counselling in primary care is widely recognized. Exercise is frequently identified as a key intervention for many chronic conditions, yet it remains under-prescribed. Physical activity counselling during routine diabetes care often takes a back seat to other issues, or lacks specific, actionable details that are important for patients to successfully integrate regular physical activity into their lifestyle. Moreover, even when prescribed, the successful implementation of physical activity behaviour changes remains a challenge for patients.

Eligible Rosemount Family Health Organization adult patients age >=18 years with type 2 diabetes mellitus will receive an email or mail invitation to self-refer to a structured, facility-based, supervised aerobic and resistance exercise program. Interested patients will be invited to attend a 1-hour information session at the exercise facility at the time of implementation start up where they will complete an initial survey. Patients will then be free to attend up to 6 regularly-scheduled, group, free classes per week at a local exercise facility for a period of 3-months. Classes will be supervised by experienced trainers.

Measures of program success will focus around four themes, informed in part by the Institute for Healthcare Improvement's Triple Aim: (i) adherence to CDA guidelines for physical activity, (ii) patient experience, and (iii) health impact. Our balancing measure will be potential costs incurred by patients. Adherence measures, including percentage uptake (i.e. attend introductory session and one class), retention (at 1, 2 and 3-months), and percentage who meet CDA recommendations for exercise will be collected. Reasons for declined or discontinued participation will also be collected voluntarily from patients to help identify concrete or perceived barriers to structured exercise programs. Health-related measures will include quality of life (EQ-5D-5L) and exercise self-efficacy (Basic Psychological Needs in Exercise Scale, BP-NES). These will be measured by patient-report at 0, 1, 2, and 3-months. Participants will be asked to rate their "willingness to recommend" (Likert scale 1-10) the program to other individuals with T2DM. Additionally, pre- and post-exercise program hemoglobin A1c and blood pressure measurements (both of which are routinely collected for all patients with T2DM) will be obtained from patient charts. Finally, while this program will be free to patients, a hypothetical cost per patient will be estimated in order to gain an understanding of the financial costs compared to the value added through patient experience and health outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >= 18 years) patients rostered with one of the Rosemount Clinic physicians with a clinical diagnosis of type 2 diabetes mellitus (fasting plasma glucose of >= 7.0 mmol/L, a 2-hour plasma glucose value in a 75 g oral glucose tolerance test of >= 11.1 mmol/L or a glycated hemoglobin (A1C) of >= 6.5%).

Exclusion Criteria:

Exclusion criteria are primarily based off of those employed in the Look AHEAD (Action for Health in Diabetes) trial. The Look AHEAD trial is the largest randomized trial to date evaluating the efficacy of a physical activity and dietary control intervention in older adults with type 2 diabetes (Espeland, M. et al. 2003. Look AHEAD [Action for Health in Diabetes]: design and methods for a clinical trial of weight loss for the prevention of cardiovascular disease in type 2 diabetes. Controlled Clinical Trials. 24:610-628.).

* Pregnant
* A1C > 11%
* Blood pressure >= 160/100 mmHg
* Fasting triglycerides >= 600 mg/dL
* Underlying diseases that may limit life span and/or affect the safety of the intervention:
* Currently pregnant or less than 3 months post-partum
* CVD event within the past 3 months (STEMI or NSTEMI)
* CVD manifesting any of the following criteria: Unstable angina pectoris or angina pectoris at rest, positive cardiac stress testing without completed work up or intervention, history of cardiac arrest, complex ventricular arrhythmia at rest or with exercise, uncontrolled atrial fibrillation (heart rate of 100 beats per minute or more), New York Heart Association Class III or IV congestive heart failure, acute myocarditis, pericarditis, hypertrophic cardiomyopathy, clinically significant aortic stenosis, cardiac pacemaker - unless approved by a Cardiologist, implantable cardioverter defribrillator (ICD) device in situ, history of aortic aneurysm of at least 7 cm in diameter or aortic aneurysm repair, resting heart rate < 45 beats per minute or > 100 beats per minute, or heart transplantation.
* Documented history of pulmonary embolus in past 6 months
* Currently undergoing active cancer treatment
* Renal disease manifesting any of the following criteria: Urine dipstick protein 4+, rerum creatinine > 124 µmol/L (female) or > 133 µmol/L (male), or currently receiving dialysis
* Untreated proliferative neuropathy
* Actively infected foot ulcer
* Chronic obstructive pulmonary disease that would limit ability to participate in intervention
* Chronic hepatitis B or C cirrhosis
* Inflammatory bowel disease requiring corticosteroid treatment for acute flare within the past year
* Endocrine disorder: Type 1 Diabetes, Cushing's syndrome or acromegaly
* Any major organ transplant
* HIV-positive
* Active tuberculosis
* Factors that may limit adherence to intervention: Inability to walk two blocks, lack of fluency in spoken English or French, hospitalization for depression in past 6 months, current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder, self-report of alcohol or substance use disorder within the past 12 months, or lack of support from Rosemount Clinic physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Program adherence | 3-months
  Percentage of participants who meet or exceed Canadian Diabetes Association guideline recommendations for exercise in type 2 diabetes
Program uptake | 3-months
  Percentage of participants who attend the introductory session and at least one group class
Program retention | 3-months
  Retention rate of participants

SECONDARY OUTCOMES:
Health-related quality of life | 0, 1, 2 and 3-months
  Change from baseline in 5-level EuroQol-5 Domain score (this is a quality of life scale where higher values indicate better quality of life) with Canadian index scores ranging from -0.148 (worst state) to 0.949 (best state).
Psychological experience with exercise | 0, 1, 2 and 3-months
  Change from baseline in Basic Psychological Needs in Exercise Scale (measuring basic psychological needs in healthy physical exercise) score with scores ranging from 11 (worst) to 55 (best) (in other words higher scores indicate that needs are better met).
Willingness to recommend | 3-months
  Participants will be asked to rate their "willingness to recommend" (Likert scale) the program to other individuals with type 2 diabetes (this is a 10-point scale where higher values indicate higher likelihood to recommend).
Blood pressure | 0 and 3-months
  Baseline and post-intervention blood pressure measurements will be obtained from patient charts, as routinely collected during type 2 diabetes care every 3-months.
Hemoglobin A1c | 0 and 3-months
  Baseline and post-intervention hemoglobin A1c measurements will be obtained from patient charts, as routinely collected during type 2 diabetes care every 3-months.
Hypothetical program cost per patient | 3-months
  A hypothetical program cost per patient will be estimated to balance against the program benefits.

IPD SHARING:
Plan to Share IPD: No